CLINICAL TRIAL: NCT02013349
Title: POST-MARKET EVALUATION OF DESolve® NOVOLIMUS ELUTING BIORESORBABLE CORONARY SCAFFOLD SYSTEM IN THE TREATMENT OF PATIENTS WITH DE NOVO NATIVE CORONARY ARTERY LESIONS
Brief Title: DESolve Post-Approval Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elixir Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELX-CL-1203
Record Dates: First submitted 2013-12-06; First posted 2013-12-17 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: prospective, multi-center registry
Oversight: Data Monitoring Committee: No

ARMS (1):
- DESyne Novolimus Eluting CSS (Other): approved device continued access
  Interventions: Device: coronary intervention

INTERVENTIONS:
Device: coronary intervention

SUMMARY:
To evaluate the long-term safety and performance of the DESolve Novolimus Eluting Bioresorbable Coronary Scaffold System

DETAILED DESCRIPTION:
DESolve is not currently approved for sale in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years of age
* Patient is able to verbally confirm understanding of risks, benefits and treatment alternatives of receiving the DESolve NE BCSS and he/she provides written informed consent, as approved by the appropriate Ethics Committee of the respective clinical site, prior to any clinical study related procedure
* Patient must have evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia, positive functional study or electrocardiogram (ECG) changes consistent with ischemia)
* Patient must be an acceptable candidate for coronary artery bypass graft (CABG) surgery
* Patient must agree to undergo all clinical study required follow-up visits
* Patient must agree not to participate in any other clinical study for a period of two years following the index procedure

Angiographic Inclusion Criteria - Target Lesion/Vessel Target lesion must be located in a native coronary artery with a nominal vessel diameter of between 2.75 and 3.5 mm assessed by visual estimation or QCA

* Target lesion must measure ≤ 24 mm in length
* Target lesion must be in a major artery or branch with a visually estimated stenosis of ≥ 50% and < 90% with a TIMI flow of ≥ 1
* Percutaneous intervention of lesions in the target vessel if:
* Not part of a clinical investigation
* ≥ 6 months prior to the study index procedure
* ≥ 9 months after the study index procedure (planned)
* Previous intervention was distal to and > 10 mm from the target lesion

Exclusion Criteria:

* Patient has a known diagnosis of acute myocardial infarction (AMI) within 72 hours preceding the index procedure and CK and CK-MB have not returned within normal limits at the time of procedure
* Patient is currently experiencing clinical symptoms consistent with AMI
* Patient requires the use of any rotablator intervention during the index procedure
* Patient has current unstable arrhythmias
* Patient has a known left ventricular ejection fraction (LVEF) < 30%
* Patient has received a heart transplant or any other organ transplant or is on a waiting list for any organ transplant
* Patient is receiving or scheduled to receive chemotherapy for malignancy within 30 days prior to or after the procedure
* Patient is receiving immunosuppression therapy and has known immunosuppressive or autoimmune disease (e.g. human immunodeficiency virus, systemic lupus erythematosus)
* Patient is receiving chronic anticoagulation therapy (e.g., heparin, Coumadin) that cannot be stopped and restarted according to local hospital standard procedures
* Patient has a known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, both clopidogrel and ticlopidine, Novolimus, PLLA polymers or contrast sensitivity that cannot be adequately pre-medicated
* Elective surgery is planned within the first 6 months after the procedure that will require discontinuing either aspirin or clopidogrel
* Patient has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3, a WBC of < 3,000 cells/mm3, or documented or suspected liver disease
* Patient has known renal insufficiency (e.g., serum creatinine level of more than 2.5 mg/dL, or patient on dialysis)
* Patient has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Patient has had a cerebrovascular accident (CVA) or transient ischemic neurological attack (TIA) within the past six months
* Patient has had a significant GI or urinary bleed within the past six months
* Patient has extensive peripheral vascular disease that precludes safe 6 French sheath insertion
* Patient has other medical illness (e.g., cancer or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the clinical study plan, confound the data interpretation or is associated with a limited life expectancy (i.e., less than one year)
* Patient is already participating in another clinical study
* Women of childbearing potential who have not undergone surgical sterilization or are not post-menopausal (defined as amenorrheic for at least one year) as well as women who are pregnant or nursing
* Patient is unable to give their consent, is legally incompetent, or is institutionalized by virtue of an order issued by the courts or other authority

Angiographic Exclusion Criteria - Target Lesion/Vessel

* Target lesion(s) meets any of the following criteria:
* Aorto-ostial location
* Left main location
* Located within 5 mm of the origin of the LAD or LCX
* Located within an arterial or saphenous vein graft or distal to a diseased arterial or saphenous vein graft
* Lesion involving a side branch >2mm in diameter or bifurcation
* Previous placement of a scaffold proximal to or within 10 mm of the target lesion
* Total occlusion (TIMI flow 0), or sub-total occlusion (TIMI flow 1)
* Excessive tortuosity proximal to or within the lesion
* Angulation (≥ 45o) proximal to or within the lesion
* Calcification moderate or heavy
* Previous intervention restenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2014-04-22 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | 1 month
  Major Adverse Cardiac Events (MACE) is defined as cardiac death, MI not clearly attributable to a non-intervention vessel, and clinically-indicated target lesion revascularization
Major Adverse Cardiac Events (MACE) | 6 months
  Major Adverse Cardiac Events (MACE) is defined as cardiac death, MI not clearly attributable to a non-intervention vessel, and clinically-indicated target lesion revascularization
Major Adverse Cardiac Events (MACE) | 12 months
  Major Adverse Cardiac Events (MACE) is defined as cardiac death, MI not clearly attributable to a non-intervention vessel, and clinically-indicated target lesion revascularization
Major Adverse Cardiac Events (MACE) | 2 years
  Major Adverse Cardiac Events (MACE) is defined as cardiac death, MI not clearly attributable to a non-intervention vessel, and clinically-indicated target lesion revascularization
Major Adverse Cardiac Events (MACE) | 3 years
  Major Adverse Cardiac Events (MACE) is defined as cardiac death, MI not clearly attributable to a non-intervention vessel, and clinically-indicated target lesion revascularization
Major Adverse Cardiac Events (MACE) | 4 years
  Major Adverse Cardiac Events (MACE) is defined as cardiac death, MI not clearly attributable to a non-intervention vessel, and clinically-indicated target lesion revascularization
Major Adverse Cardiac Events (MACE) | 5 years
  Major Adverse Cardiac Events (MACE) is defined as cardiac death, MI not clearly attributable to a non-intervention vessel, and clinically-indicated target lesion revascularization

CONTACTS AND LOCATIONS:
Locations (7):
- Germany (4):
  - Herz-Kreislaufzentrum Bad Segeberg, Bad Segeberg
  - Universitätsklinikum Giessen und Marburg GmbH, Giessen
  - Universitätsklinikum Münster, Münster
  - Krankenhaus der Barmherzigen Brüder, Trier
- Ospendale San Raffaele, Milan, Italy
- Jordan (2):
  - Jordan Hospital, Amman
  - King Abdullah University Hospital, Irbid